CLINICAL TRIAL: NCT05723536
Title: PLAI-AF Trial: Hybrid Endo-epicardial Partial Left Atrial Isolation vs. Endocardial Ablation in Patients With Persistent Atrial Fibrillation
Acronym: PLAI-AF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2022/1059
Record Dates: First submitted 2023-02-02; First posted 2023-02-10 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation; Persistent Atrial Fibrillation; Arrythmia
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: 1:1 randomized clinical trial in patients with persistent and long-standing persistent AF in two groups: conventional ablation vs partial endo-epicardial isolation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PLAI (Partial Left Atrial Isolation) (Experimental): Partial electrical isolation of the left atrium endo-epicardially (pulmonary veins, posterior wall and left atrial appendage) and left atrial appendage isolation using Atriclip (Atricure, Mason OH, USA) in a single procedure in patients with persistent atrial fibrillation.
  Interventions: Procedure: Partial Left Atrial Isolation
- CA (Catheter Ablation) (Active Comparator): Conventional catheter ablation of persistent atrial fibrillation.
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Procedure: Partial Left Atrial Isolation — Partial electrical isolation of the left atrium endo-epicardially (pulmonary veins, posterior wall and left atrial appendage) and left atrial appendage isolation using Atriclip (Atricure, Mason OH, USA) in a single procedure in patients with persistent atrial fibrillation.
  Arms: PLAI (Partial Left Atrial Isolation)
Procedure: Catheter Ablation — Catheter Ablation of Atrial Fibrillation
  Arms: CA (Catheter Ablation)

SUMMARY:
In patients with symptomatic atrial fibrillation (AF), current clinical guidelines recommend ablation for rhythm control.

While percutaneous ablation has good results in patients with paroxysmal AF, it is not clear which is the best technique in patients with persistent or long-standing persistent AF. Our group performed the first randomized study of thoracoscopic epicardial ablation vs. endocardial catheter ablation (FAST Trial), which showed better results for epicardial ablation but with a higher rate of complications. Hybrid epicardial and endocardial ablation strategies have recently been described sequentially, showing better results in patients with persistent AF, but 40% of patients are still refractory to ablation.

Our study aims to compare the conventional strategy (catheter ablation) with partial electrical isolation of the left atrium endo-epicardially (pulmonary veins, posterior wall and left atrial appendage) in a single procedure in the group of patients most refractory to ablation. Likewise, using magnetic resonance imaging and echocardiography to analyze the atrial remodeling factors that can predict the success and failure of both therapies.

Methodology: A 1:1 randomized clinical trial in patients with persistent and long-standing persistent AF in two groups: conventional ablation vs. partial endo-epicardial isolation. Prior to ablation, cardioversion will be performed and functionality and atrial size will be verified by echocardiography and delayed-enhancement magnetic resonance imaging (MRI) will detect the degree of fibrosis and atrial remodeling. During the ablation procedure, a continuous rhythm recording device will be implanted. Likewise, at three months the MRI will be repeated to detect post-ablation fibrosis. At six months the echocardiography will be performed to assess atrial function and size.

Main Expected Results: The expected results include: 1. an improvement in the rate of patients with no atrial arrhythmias recurrence in patients undergoing endo-epicardial ablation; 2. a lower AF burden in patients undergoing endo-epicardial ablation who have had recurrence; 3. To know the degree of atrial fibrosis associated with the success/failure of each technique; 4. To know the degree of fibrosis that both techniques produce; 5. To know the degree of ventricular function associated with the success/failure of each technique; 6. To know the degree of potentially lost atrial function; 7. To Compare the safety of both techniques

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18 and 75, both inclusive, at the time of the consent date.
2. Patients with persistent atrial fibrillation refractory to at least one antiarrhythmic drug (Class I or III).
3. Signature of written informed consent.

Exclusion Criteria:

1. Persistent atrial fibrillation of more than 4 years.
2. Moderate to severe valvular heart disease.
3. Severe atrial dilatation (left appendage AP diameter > 55 mm or > 50ml/m2).
4. Patients requiring concomitant cardiac surgery or with previous cardiac surgery.
5. Left ventricular ejection fraction <40%.
6. History of pericarditis.
7. Previous stroke.
8. Presence of active infection or sepsis, esophageal ulcer stricture and/or esophageal varices.
9. Patients with renal dysfunction defined as GFR less than or equal to 40 ml/min/m2.
10. Contraindication for chronic anticoagulation.
11. Patients who have undergone prior left atrial catheter ablation for atrial fibrillation or who are receiving treatment for ventricular arrhythmia.
12. Patients with severe chronic obstructive pulmonary disease considered GOLD III.
13. Patients with active neoproliferative disease or other concomitant disease where the medical team considers that ablation places the patient at unacceptable risk.
14. Pregnant, lactating women.
15. Patients who have previously presented allergic reactions to gadolinium.
16. Patients with claustrophobia that makes it impossible to perform nuclear magnetic resonance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Absence of atrial arrhythmia | 3-12 months post-surgery
  Success or failure to be free of atrial arrhythmias (AF/AT/AFL) in the absence of class I and III antiarrhythmic drugs, or with the same antiarrhythmic treatment prior to study inclusion, after the 3-month blank period, during 12 months after the procedure and measured by loop recorder.

SECONDARY OUTCOMES:
90% reduction in baseline AF burden | 3-12 months post-surgery
  90% reduction in baseline AF burden in the absence of a new/increased dose of class I/III antiarrhythmic medication, as measured by implantable ECG recorder.
Pre-procedure atrial remodeling | 3-months pre-surgery to 12 months post-surgery
  Pre-procedure atrial remodelling by MRI measuring fibrosis grade. Pre-procedure atrial remodelling by echocardiogram measuring size and function. Both measurements are in relation to primary endpoint success/failure in both groups.
Post-procedure atrial remodeling | 3-12 months post-surgery
  Post-procedure atrial remodelling by MRI measuring fibrosis grade. Post-procedure atrial remodelling by echocardiogram measuring size and function. Both measurements are in relation to primary endpoint success/failure in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Background] Castella M, Kotecha D, van Laar C, Wintgens L, Castillo Y, Kelder J, Aragon D, Nunez M, Sandoval E, Casellas A, Mont L, van Boven WJ, Boersma LVA, van Putte BP. Thoracoscopic vs. catheter ablation for atrial fibrillation: long-term follow-up of the FAST randomized trial. Europace. 2019 May 1;21(5):746-753. doi: 10.1093/europace/euy325. PMID 30715255
- [Background] Boersma LV, Castella M, van Boven W, Berruezo A, Yilmaz A, Nadal M, Sandoval E, Calvo N, Brugada J, Kelder J, Wijffels M, Mont L. Atrial fibrillation catheter ablation versus surgical ablation treatment (FAST): a 2-center randomized clinical trial. Circulation. 2012 Jan 3;125(1):23-30. doi: 10.1161/CIRCULATIONAHA.111.074047. Epub 2011 Nov 14. PMID 22082673
- [Background] Maesen B, Pison L, Vroomen M, Luermans JG, Vernooy K, Maessen JG, Crijns HJ, La Meir M. Three-year follow-up of hybrid ablation for atrial fibrillation. Eur J Cardiothorac Surg. 2018 Apr 1;53(suppl_1):i26-i32. doi: 10.1093/ejcts/ezy117. PMID 29590387
- [Background] DeLurgio DB, Crossen KJ, Gill J, Blauth C, Oza SR, Magnano AR, Mostovych MA, Halkos ME, Tschopp DR, Kerendi F, Taigen TL, Shults CC, Shah MH, Rajendra AB, Osorio J, Silver JS, Hook BG, Gilligan DM, Calkins H. Hybrid Convergent Procedure for the Treatment of Persistent and Long-Standing Persistent Atrial Fibrillation: Results of CONVERGE Clinical Trial. Circ Arrhythm Electrophysiol. 2020 Dec;13(12):e009288. doi: 10.1161/CIRCEP.120.009288. Epub 2020 Nov 13. PMID 33185144
- [Background] Yorgun H, Canpolat U, Kocyigit D, Coteli C, Evranos B, Aytemir K. Left atrial appendage isolation in addition to pulmonary vein isolation in persistent atrial fibrillation: one-year clinical outcome after cryoballoon-based ablation. Europace. 2017 May 1;19(5):758-768. doi: 10.1093/europace/eux005. PMID 28340073
- [Background] Whitlock RP, Belley-Cote EP, Paparella D, Healey JS, Brady K, Sharma M, Reents W, Budera P, Baddour AJ, Fila P, Devereaux PJ, Bogachev-Prokophiev A, Boening A, Teoh KHT, Tagarakis GI, Slaughter MS, Royse AG, McGuinness S, Alings M, Punjabi PP, Mazer CD, Folkeringa RJ, Colli A, Avezum A, Nakamya J, Balasubramanian K, Vincent J, Voisine P, Lamy A, Yusuf S, Connolly SJ; LAAOS III Investigators. Left Atrial Appendage Occlusion during Cardiac Surgery to Prevent Stroke. N Engl J Med. 2021 Jun 3;384(22):2081-2091. doi: 10.1056/NEJMoa2101897. Epub 2021 May 15. PMID 33999547
- [Background] Bisbal F, Benito E, Teis A, Alarcon F, Sarrias A, Caixal G, Villuendas R, Garre P, Soto N, Cozzari J, Guasch E, Junca G, Prat-Gonzalez S, Perea RJ, Bazan V, Tolosana JM, Arbelo E, Bayes-Genis A, Mont L. Magnetic Resonance Imaging-Guided Fibrosis Ablation for the Treatment of Atrial Fibrillation: The ALICIA Trial. Circ Arrhythm Electrophysiol. 2020 Nov;13(11):e008707. doi: 10.1161/CIRCEP.120.008707. Epub 2020 Oct 8. PMID 33031713
- [Background] Bisbal F, Guiu E, Cabanas-Grandio P, Berruezo A, Prat-Gonzalez S, Vidal B, Garrido C, Andreu D, Fernandez-Armenta J, Tolosana JM, Arbelo E, de Caralt TM, Perea RJ, Brugada J, Mont L. CMR-guided approach to localize and ablate gaps in repeat AF ablation procedure. JACC Cardiovasc Imaging. 2014 Jul;7(7):653-63. doi: 10.1016/j.jcmg.2014.01.014. Epub 2014 May 7. PMID 24813966
- [Background] Althoff TF, Garre P, Caixal G, Perea R, Prat S, Tolosana JM, Guasch E, Roca-Luque I, Arbelo E, Sitges M, Brugada J, Mont L. Late gadolinium enhancement-MRI determines definite lesion formation most accurately at 3 months post ablation compared to later time points. Pacing Clin Electrophysiol. 2022 Jan;45(1):72-82. doi: 10.1111/pace.14415. Epub 2021 Dec 15. PMID 34820857
- [Background] Sanz-de la Garza M, Grazioli G, Bijnens BH, Sarvari SI, Guasch E, Pajuelo C, Brotons D, Subirats E, Brugada R, Roca E, Sitges M. Acute, Exercise Dose-Dependent Impairment in Atrial Performance During an Endurance Race: 2D Ultrasound Speckle-Tracking Strain Analysis. JACC Cardiovasc Imaging. 2016 Dec;9(12):1380-1388. doi: 10.1016/j.jcmg.2016.03.016. Epub 2016 Aug 17. PMID 27544898
- [Background] Gabrielli L, Herrera S, Contreras-Briceno F, Vega J, Ocaranza MP, Yanez F, Fernandez R, Saavedra R, Sitges M, Garcia L, Chiong M, Lavandero S, Castro PF. Increased active phase atrial contraction is related to marathon runner performance. Eur J Appl Physiol. 2018 Sep;118(9):1931-1939. doi: 10.1007/s00421-018-3927-7. Epub 2018 Jul 3. PMID 29971492